CLINICAL TRIAL: NCT00498849
Title: The Changes of Patterns of Microarray in Patients With Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9361701236; NSC 94-2314-B-002-218-
Record Dates: First submitted 2007-07-08; First posted 2007-07-10 (Estimated); Last update posted 2007-07-10 (Estimated); Status verified 2005-01

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Sleep apnea; Continuous positive airway pressure; Microarray; Polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CPAP

SUMMARY:
The aim of this study are (1) To genome-wide profile the gene expression patterns of peripheral blood mononuclear cell (PBMC) in patients with obstructive sleep apnea (OSA) (2) To profile the gene expression patterns change before and after treatment with continuous positive airway pressure (CPAP) (3) To correlate the altered gene expression with the severity of the disease and outcome of OSA patients

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) is characterized with recurrent collapse of upper airway during sleep and resulted in hypoxia and sleep fragmentation. Several systemic and cardiovascular complications have been attributed to OSAS, which is caused by hypoxia and bursts of sympathetic activity. Increase of inflammatory mediators, which included C-reactive protein, oxidative stress, adhesion molecules, vascular endothelial growth factor and proinflammatory cytokines, were thought to involve in the developments of cardiovascular diseases in patients with OSAS. In our preliminary study, both serum levels of IL-6 and CRP were higher in patients with OSAS than control subjects, and the levels were inversely correlated with the lowest pulse oxygen saturation. Factors triggering inflammatory cascades in OSAS included hypoxia and sympathetic hyperactivity.

Hypoxia was thought to be the trigger factor for the elevated production of inflammatory mediators. Through the induction of transcriptional factors and critical signaling pathways, hypoxia induces several physiologic responses, like increased anaerobic metabolism, angiogenesis, vasodilation, erythropoiesis and increased breathing.

Microarray is the more mature gene analysis techniques so far, which can allow high throughput analysis of the function of many genes. Microarray can be used to understand the disease mechanisms and is also very useful to improve disease diagnosis, disease classification, prognosis evaluation and to improve treatment outcome. In this project, we use oligo microarray to genome-wide profile the altered gene expressions in peripheral blood mononuclear cells of OSAS patients; and to correlate the dysregulations of gene expression with the clinical outcome. We will also examine the gene expression patterns change before and after treatment with CPAP. The information obtained by this approach will be very useful to understand the pathogenic mechanism of OSAS that leads to the systemic and cardiovascular complications. Further therapeutic intervention may therefore be possible.

ELIGIBILITY:
Inclusion Criteria:

* healthy control with age > 18 y/o severe OSA (AHI>=30/hr) with age>18 y/o

Exclusion Criteria:

* chronic lung disease female refuse to receive CPAP treatment or poor compliant to CPAP neurologic event

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-02; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
CPAP effect | 4-week after CPAP treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peilin Lee, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- Naitonal Taiwan Univerisity Hospital, Taipei, Taiwan